CLINICAL TRIAL: NCT00280319
Title: Randomized Controlled Study of Non-pharmacologic Treatments for Depression Among Displaced Adolescents in Northern Uganda.
Brief Title: Study of Treatments for Depression Among Displaced Adolescents in Northern Uganda.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: World Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BUWVRCT2
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Depression
Keywords: randomized controlled trial; depression; Uganda; adolescents
MeSH Terms: conditions — Depression | interventions — Interpersonal Psychotherapy; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IPT arm (Experimental): interpersonal psychotherapy for groups (IPT-G). this consists of psychotherapy provided to participants in a group format.
  Interventions: Behavioral: interpersonal psychotherapy for groups
- CP arm (Experimental): Creative Play therapy consists of play activities provided to participants in groups.
  Interventions: Behavioral: creative play therapy
- control (No Intervention): those who are wait-list controls

INTERVENTIONS:
Behavioral: interpersonal psychotherapy for groups — psychotherapy
  Arms: IPT arm
Behavioral: creative play therapy — consisted of play activities
  Arms: CP arm

SUMMARY:
That interpersonal psychotherapy and creative play therapies can reduce symptoms of depression among adolescents with depressive-type illness in northern Uganda.

DETAILED DESCRIPTION:
This study represents the third phase of a project aimed at developing, validating, and using locally-relevant assessments of emotional and behavioral problems in Acholi war-affected children to evaluate interventions being delivered by non-governmental organizations in the N. of Uganda. It is positioned to make a unique contribution to the field by both developing culturally appropriate screening and assessment methods and then using them to assess the efficacy of an adapted, manualized treatment both pre-and post-intervention.

The intent of the proposed intervention study is to test the efficacy of group interpersonal psychotherapy (IPT) for treatment of specific psychosocial problems and associated impairment in Acholi IDP adolescents living in the Unyama and Awer camps of Gulu District, Northern Uganda. These interventions represent the existing standard of care provided by NGOs working in this region, but. for tje first time, collaboration of the NGOs in this study will help ensure systematic assessment of participants to investigate the efficacy of interventions being offered.

The proposed research study aims to test the efficacy of a group treatment for emotional and behavioral problems in war-affected adolescents. Emotional and behavioral problems will be assessed using a locally-validated scale of psychosocial problems and functional impairment developed from ethnographic work conducted in the same IDP camps in Gulu District in July 2004. The intervention to be tested will be group interpersonal therapy (IPT) which has shown efficacy for use in treating depression in Ugandan adults In Masaka and Rakai provinces. The decision to use IPT in this IDP population was based on the fact that symptoms similar to depression and comorbid anxiety, for which IPT is indicated, dominated in the ethnographic assessment of emotional and behavioral problems collected in July. Additionally, we have prior direct experience in Uganda that IPT can be easily trained and systematically delivered in a low-resource environment lay practitioners and that it is effective in treating depression. Furthermore, our ethnographic work has resulted in a suitable measure for assessing emotional and behavioral problems in war- affected Acholi youth living in the Northern Uganda for use in screening adolescents into intervention groups. The application of valid instruments to assess psychosocial problems and the degree of impairment both pre and post- intervention will be invaluable to our implementing partners - World Vision/War Child - for developing effective interventions to address the ongoing mental health needs of the young people they serve in Northern Uganda.

Specific Objectives 1. To assess symptoms of locally described depression-like syndromes (Kumu/Par/Two Tam), a local anxiety syndrome (Ma Lwor) and social problems (Gin lugero/tic marac) in Acholi war-affected adolescents using the Acholi Psychosocial Assessment Instrument (APAI), a locally-derived tool for assessment of emotional and behavioral problems in children and youth available in the Luo language.

2. To randomly assign screened individuals found to have these problems to one of three treatment conditions including: a) group IPT; b) a facilitated arts & recreation control condition; and c) a wait-list control condition.

3. To conduct post-intervention testing and comparison of all treatment conditions using the APAI. This will be done immediately after the IPT intervention is completed, and repeated 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* aged 14-17 years. living in displaced persons camps in northern Uganda meet study-specific criteria for depression

Exclusion Criteria:

* reported age of less than 14 or older than 17 years does not live in a displaced persons camp

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 338 (Actual)
Dates: Start 2005-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
depression | pre, post and 6 months post treatment
  adapted depression instrument - HSCL.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bolton, MB BS, Principal Investigator — Boston University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bolton P, Bass J, Betancourt T, Speelman L, Onyango G, Clougherty KF, Neugebauer R, Murray L, Verdeli H. Interventions for depression symptoms among adolescent survivors of war and displacement in northern Uganda: a randomized controlled trial. JAMA. 2007 Aug 1;298(5):519-27. doi: 10.1001/jama.298.5.519. PMID 17666672